CLINICAL TRIAL: NCT05460481
Title: Anlotinib Plus Penpulimab in Advanced Non-Small-Cell Lung Cancer Previously Treated With PD-1/PD-L1 Inhibitors: A Multicenter, Single-arm, Explorative Trial
Brief Title: Anlotinib Plus Penpulimab in Advanced Non-Small-Cell Lung Cancer Previously Treated With PD-1/PD-L1 Inhibitors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: Henan Cancer Hospital (Other Government); Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L045
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib; penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Anlotinib Plus Penpulimab (Experimental): Anlotinib (10mg qd po d1-14, 21 days per cycle) and Penpulimab (200mg ivgtt d1)
  Interventions: Drug: Anlotinib Plus Penpulimab

INTERVENTIONS:
Drug: Anlotinib Plus Penpulimab — Anlotinib: 10mg orally daily on day 1 to 14 of a 21-day cycle. Penpulimab: 200mg by intravenous drip on day 1 of a 21-day cycle.
  Other Names: Anlotinib & Penpulimab

SUMMARY:
Anlotinib is a multi-target receptor tyrosine kinase inhibitor in domestic research and development. It can inhibit the angiogenesis related kinase, such as VEGFR, FGFR, PDGFR, and tumor cell proliferation related kinase -c-Kit kinase. In the phase # study, patients who failed at least two kinds of systemic chemotherapy (third line or beyond) or drug intolerance were treated with anlotinib or placebo, the anlotinib group PFS and OS were 5.37 months and 9.63 months, the placebo group PFS and OS were 1.4 months and 6.3 months. Therefore, the combination of Anlotinib and Penpulimab (a new PD-1 inhibitor) is attempted for the treatment of advanced non-small-cell lung cancer (NSCLC) participants who have progressed following prior PD-1 or PD-L1 Inhibitors treatment, to further improve the patient's PFS or OS.

DETAILED DESCRIPTION:
This is a multicenter, single-arm, explorative clinical trial conducted in China to investigate the efficacy and safety of anlotinib plus docetaxel in advanced NSCLC patients (pts) who have progressed following prior PD-1 or PD-L1 Inhibitors treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Non Small cell lung cancer pathologically confirmed, with measurable nidus (RECIST 1.1)
* Disease progression following prior Immune Checkpoint Inhibitors (PD-1 or PD-L1 inhibitors) treatment for NSCLC for at least 2 consecutive treatment cycles.
* EGFR/ALK/ROS1 wild type
* ECOG PS: 0-1, Expected Survival Time: Over 3 months
* Adequate bone marrow, liver and renal function
* The woman patients of childbearing age who must agree to take contraceptive methods (e.g. intrauterine device, contraceptive pill or condom) during the research and within another 8 weeks after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; The man patients who must agree to take contraceptive methods during the research and within another 8 weeks after it.

Exclusion Criteria:

* Small Cell Lung Cancer (including small cell cancer and other kinds of cancer mixed with non small cell cancer)
* Have used Anlotinib or other antiangiogenic drugs before
* Known primary multidrug resistance to prior ICIs treatments
* Have failed for two times or beyond of platinum two drugs chemotherapy (except adjunctive chemotherapy, neoadjuvant therapy and concurrent chemoradiotherapy
* Iconography (CT or MRI) shows obvious lung empty or necrotic tumor iconography (CT or MRI) shows that the tumor vessels have 5 mm or less, or Cardiovascular involvement by Central tumor; Or obvious lung empty or necrotic tumor
* Patients with brain or central nervous system metastases, including leptomeningeal disease, or CT/MRI examination revealed brain or leptomeningeal disease） (28 days before the random treatment has been completed and the symptoms of patients with brain metastases from stable can into the group, but need to the cerebral MRI, CT or vein angiography confirmed as without symptoms of cerebral hemorrhage)
* Patients are participating in other clinical studies (other than non-interventional studies) less than 4 weeks from the end of the previous clinical study
* Patients who had received chemotherapy, radiation, or other experimental anticancer therapy (except Diphosphonate) within 4 weeks prior to the first dose of this study. Those who had previously received local radiotherapy were eligible if they met the following criteria: the end of radiotherapy was more than 4 weeks from the start of this study (brain radiotherapy was more than 2 weeks); In addition, the target lesions selected in this study were not in the radiotherapy area, or if the target lesion is within the radiotherapy area but progression has been confirmed
* Other kinds of malignancies within 5 years or for now
* Patients who have an active, known or suspected autoimmune disease, including a history of allogeneic organ transplantation, allogeneic hematopoietic stem cell transplantation, a history of being HIV positive, or a history of acquired immunodeficiency syndrome (AIDS)
* Active or previously recorded inflammatory bowel disease (such as Crohn's disease, ulcerative colitis)
* Have got non remissive toxic reactions derived from previous therapies, which is over level 1 in CTC AE (4.0), alopecia NOT included
* Abnormal coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT ULN > 1.5), with bleeding tendency or be treated with thrombolysis and anticoagulation
* Have clinical significant hemoptysis occurred within 3 months before enrollment (daily hemoptysis more than half tablespoonl; Or clinical significant bleeding symptoms or bleeding tendency in the 4 weeks prior to grouping, such as gastrointestinal bleeding, hemorrhagic gastric ulcer (including gastrointestinal perforation and/or fistula, but gastrointestinal perforation or fistula has been surgically removed, admission is allowed), baseline fecal occulted blood ++ or above, unhealed wounds, ulcers or fractures, etc
* Urine routines show urine protein≥ ++, and urine protein quantity≥ 1.0 g during 24 hours
* Uncontrollable hypertensive (SBP≥ 150 mmHg, DBP≥100 mmHg, despite the best drug treatment)
* Patients with severe cardiovascular disease: grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmia; According to NYHA standard, grade III to IV cardiac insufficiency, or echocardiography indicates left ventricular ejection fraction (LVEF) < 50%;
* Patients with NCI-CTCAE grade II or greater peripheral neuropathy, except due to trauma
* Interstitial lung disease, uncontrolled medium to large serosal effusion (including pleural effusion, ascites, and pericardial effusion) after pumping treatment, aggravated chronic obstructive pulmonary disease, active pulmonary infection and/or acute bacterial or fungal respiratory disease requiring intravenous antibiotic treatment within 28 days
* Have an obvious factor influencing oral drug absorption, such as unable to swallow, chronic diarrhea and intestinal obstruction, etc
* Have venous thromboembolism events within 6 months before enrollment, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc
* Have received live or attenuated vaccine within 30 days prior to the initial administration of Penpulimab, or was scheduled to receive live or attenuated vaccine during the study
* Patients who have known a history of severe hypersensitivity to other monoclonal antibodies
* Patients who have known a history of psychotropic substance abuse, alcohol abuse, or drug abuse
* Uncontrolled active hepatitis after treatment (hepatitis b: HBsAg positive and HBV DNA more than 1 x 104 copy /ml; Hepatitis c: HCV RNA is positive and liver function is abnormal); Combined with hepatitis b and hepatitis c infection
* Serious diseases that endanger patients' safety or affect patients' completion of research, according to the researchers' judgment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2022-06-12 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to approximately 24 months
  Objective Response Rate per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Progress free survival (PFS) | up to approximately 24 months
  Progress free survival per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Overall Survival (OS) | up to approximately 24 months
  Overall Survival per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Disease Control Rate (DCR) | up to approximately 24 months
  Disease Control Rate per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
Safety | From the first assignment of informed consent form up to 21 days after the last dose
  Safety as measured by the rate of AEs, SAEs and laboratory abnormalities

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external indepentent Review Panel. Requestors will be required to sign a Data Access Agreement.